CLINICAL TRIAL: NCT06784791
Title: Preoperative Amivantamab or Amivantamab and Carboplatin/Pemetrexed Treatment in Patients With Resectable Non-small-cell Lung Cancer Harboring Oncogenic EGFR Mutations (NEOpredict-EGFR)
Acronym: NEOpredict-EGF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEOpredict-EGFR; 2023-505662-28-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-04; First posted 2025-01-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (NSCLC)
Keywords: NSCLC; Lung cancer; non-small-cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Carboplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Multicenter, international, open-label, two-stage design, non-randomized
Masking Description: Open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-operative amivantamab monotherapy (Experimental): Patients in stage 1 will receive 1 cycle (28 days) of pre-operative amivantamab monotherapy, splitted on 5 treatment days. Dosing will be weight-adapted.
  Interventions: Drug: Amivantamab Intravenous
- Amivantamab + chemotherapy (Experimental): Patients in stage 2 will receive 1 cycle (28 days) of pre-operative amivantamab monotherapy, splitted on 5 treatment days (dosing will be weight-adapted) plus additional chemotherapy (carboplatin/pemetrexed) on day 1.
  Interventions: Drug: Amivantamab Intravenous; Drug: Carboplatin/Pemetrexed

INTERVENTIONS:
Drug: Amivantamab Intravenous — Stage 1: Pre-operative amivantamab monotherapy Stage 2: Pre-operative amivantamab treatment plus chemotherapy (carboplatin/pemetrexed)
  Other Names: Chemotherapy
Drug: Carboplatin/Pemetrexed — Stage 2: Pre-operative amivantamab plus chemotherapy (carboplatin/pemetrexed)
  Arms: Amivantamab + chemotherapy

SUMMARY:
The primary objective of this study is to determine the feasibility of four weeks of preoperative antibody therapy with amivantamab. Amivantamab will be administered as monotherapy (stage 1), and combined with carboplatin/pemetrexed chemotherapy (stage 2). Study treatment is followed by standard of care surgery, and (if clinically indicated) standard of care adjuvant therapy (chemotherapy, radiotherapy, EGFR tyrosine kinase inhibitor therapy) in patients with early stage or locally advanced non-small-cell lung cancer harboring oncogenic EGFR mutations who are eligible for curative resection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically (core biopsy) or cytologically (e.g., bronchoscopy-guided biopsy) confirmed non-small-cell lung cancer (NSCLC) eligible for anatomic resection, with the following specifications:

   * Clinical stages I B, II or selected stage III A (T3 N1, T4 with satellite nodule in the same lung N0/N1, selected T1a-T2b N2 cases considered suitable for primary surgical approach by the multidisciplinary tumor board) according to UICC 8th edition
   * Confirmation of an oncogenic EGFR mutation (EGFR p.L858R, EGFR exon 19 in-frame deletion, EGFR exon 20 in-frame insertions, EGFR p.S768I, EGFR p.L861Q, EGFR p.G719x - additional EGFR mutations with clinically validated oncogenicity and susceptibility to amivantamab may be eligible following discussion and approval by the coordinating investigator in his capacity as sponsor representative) by validated assaytechnology (e.g., diagnostic NGS or PCR-based genotyping, adhering to quality standards defined by the nNGM Lung Cancer biomarker standard operating procedure (version 007 or higher) in Germany, or equivalent in Belgium and the Netherlands) in a pretreatment biopsy (primary tumor or lymph node metastasis)
2. Males and females, ages >= 18 years, inclusive

   * A participant of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study treatment and must agree to further serum or urine pregnancy testing during the study.
   * A participant must be (as defined in Appendix IV: Contraceptive Guidance and Collection of Pregnancy Information) either of the following:

     * Not of childbearing potential
     * Of child-bearing potential and practicing true abstinence during the entire period of the study, including up to 6 months after the last dose of study treatment is given
     * Of childbearing potential and practicing 2 methods of contraception, including 1 highly effective user independent method and a second method (examples of highly effective methods of contraception are located in Appendix IV: Contraceptive Guidance and Collection of Pregnancy Information).Participant must agree to continue contraception throughout the study and through 6 months after the last dose of study treatment.
     * Note: If the childbearing potential changes after start of the study (e.g., participant of childbearing potential who is not heterosexually active becomes active, premenarchal participant experiences menarche) the participant must begin birth control, as described above
   * A participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study treatment.
   * A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 6 months after receiving the last dose of study treatment. A participant who is sexually active with a partner of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and their partner must also be practicing a highly effective method of contraception (i.e., established use of oral, injected, or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]). If the participant is vasectomized, they must still use a condom (with or without spermicide) for prevention of passage of exposure through ejaculation, but their partner is not required to use contraception.
   * A participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment.
   * Participant must be willing and able to adhere to the lifestyle restrictions specified in this protocol.
3. ECOG performance status ≤ 1
4. Exclusion of extensive mediastinal lymph node metastases (multilevel N2, N3) by PET/CT and/or invasive mediastinal lymph node staging by EBUS-TBNA and/or staging mediastinoscopy as performed by institutional guidelines.
5. Exclusion of distant metastases by standard of care imaging studies, which include but are not limited to PET/CT or PET/MRI, or CT or MRI of thorax, abdomen including pelvic region, and bone scan. Asymptomatic brain metastases will be excluded by MRI or contrastenhanced CT as indicated by institutional guidelines and patient factors.
6. Measurable target tumor (pre RECIST 1.1) prior to preoperative study therapy using standard imaging techniques.
7. Sufficient pulmonary function (ppFEV1>30%, ppDLCO>30%) to undergo curative lung cancer surgery. Exercise tests should be performed in all patients with FEV1 or DLCO <60% of normal. In case of cardiopulmonary exercise testing, the following basic cut-off values for VO2-peak should be considered: >75% predicted or >20 mL·kg-1·min-1 qualify for pneumonectomy; <35% predicted or <10 mL·kg-1·min-1 indicate high risk for any resection. There is insufficient evidence to recommend specific cut-off values for lobectomy or segmentectomy.
8. Adequate hematological, hepatic and renal function parameters:

   * Leukocytes ≥ 2,000/mm³, platelets ≥ 100,000/mm³, absolute neutrophil count (ANC) ≥ 1,500/μL, hemoglobin ≥ 9 g/dL (stage 1) or 10 g/dL (stage 2)
   * Anti-platelet therapy (such as but not limited to clopidogrel) should be discontinued pre-operatively according to local standards. If this therapy cannot be interrupted due to severe cardiovascular comorbidity, patient is ineligible for the trial
   * Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the upper limit of normal (ULN) (unless receiving anticoagulation therapy). Patients receiving warfarin/phenprocoumon or direct oral anticoagulants are to be bridged according to local standards and have achieved stable coagulation profile prior to surgery
   * Serum creatinine ≤ 1.5 x upper limit of normal and creatinine clearance >45 mL/min as measured or calculated by Cockcroft- Gault formula for estimated creatinine clearance (Appendix VII)
   * Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.0 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal. Subjects with Gilbert's syndrome can be enrolled if conjugated bilirubin is within normal limits
9. Sufficient cardiac left ventricular defined as LVEF ≥ 50% documented either by echocardiography or MUGA (echocardiography preferred, MUGA not used in German sites) within 6 months before first administration of study drug.
10. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures.

Exclusion Criteria:

1. Lung cancer entity and stage other than defined by the inclusion criteria.
2. Absence of a predictive oncogenic EGFR mutation (EGFR p.L858R, EGFR exon 19 in-frame deletion, EGFR exon 20 in-frame insertions, EGFR p.S768I, EGFR p.L861Q, EGFR p.G719x - additional EGFR mutations with clinically validated oncogenicity and susceptibility to amivantamab may be eligible following discussion and approval by the coordinating investigator in his capacity as sponsor representative) in apretreatment biopsy (primary tumor or metastasis).
3. Active or past medical history of interstitial lung disease (ILD)/pneumonitis, including drug- or radiation-induced ILD/pneumonitis.
4. Subjects with a condition requiring continuous systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted.
5. Subjects who have undergone organ transplant or allogeneic stem cell transplantation.
6. ppFEV1<30%, ppDLCO<30%, ppVO2max < 10 ml/min/kg or other criteria of functional inoperability per local guidelines.
7. History of uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

   * Myocardial infarction (MI), NSTEMI, coronary artery bypass grafting, or stroke/transient ischemic attack (TIA) within the 6 months prior to consent
   * Uncontrolled angina within the 3 months prior to consent
   * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
   * Prolonged corrected QTc interval by Fridericia's > 470 msec
   * Uncontrolled persistent hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg)
   * Clinically significant deep vein thrombosis or pulmonary embolism within 1 month prior to study treatment (clinically nonsignificant thrombosis or incidental, asymptomatic pulmonary embolism are not exclusionary)
   * Pulmonary hypertension (sPAP >35 mmHg; only measured if clinically indicated and/or mandated per local guidelines)
8. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion etc.).
9. Cardiovascular or pulmonary disease-related requirement for daily supplemental oxygen.
10. History of two or more myocardial infarctions or two or more coronary revascularization procedures.
11. Patients with active neurological disease should be excluded.
12. Active malignancy or a prior malignancy within the past 3 years. Patients with the following conditions are not excluded from participation:

    o Patients with adequately resected skin cancer (melanoma or non-melanoma), cervical carcinoma in-situ, intestinal polyps not containing invasive cancer, treated breast carcinoma in-situ or bladder carcinoma in-situ that are considered completely cured, and patients with isolated elevation in prostate-specific antigen or low risk prostate cancer managed with active surveillance or watchful waiting in the absence of radiographic evidence of metastatic prostate cancer.
13. Known history of positive test for human immunodeficiency virus (HIV- 1 and HIV-2) or known acquired immunodeficiency syndrome (AIDS). NOTE: Testing for HIV-1 and HIV-2 must be performed at screening.
14. Positive test result for hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg).

    o Note: participants with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at screening (i) a negative HBsAg and (ii) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.
15. Positive hepatitis C antibody (anti-HCV).

    o Note: participants with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
16. History of other clinically active infectious liver disease
17. Uncontrolled diabetes mellitus
18. Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment] or diagnosed or suspected viral infection.
19. Psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements.
20. Any ophthalmologic condition that is clinically unstable.
21. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of amivantamab, carboplatin or pemetrexed, or may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
22. Receipt of live attenuated vaccine within 30 days prior to the first dose of study medication.
23. Serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment
24. The patient has undergone major surgery within 28 days prior to enrollment except staging mediastinoscopy, diagnostic VATS or implantation of a venous port-system, or has not recovered from prior surgery.
25. Any other concurrent preoperative antineoplastic treatment including irradiation
26. Pregnant women
27. Breastfeeding women
28. Insufficient cardiac left ventricular function defined as LVEF<50% by echocardiography (outside Germany: or MUGA scan)
29. A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent
30. Subjects with history of severe or life-threatining (grade 3 or 4) infusion-related reactions to prior antibody therapy or immune therapy
31. Prior treatment with amivantamab or any EGFR tyrosine kinase inhibitor
32. Participation in another interventional clinical study within the last 3 months prior to inclusion or simultaneous participation in other interventional clinical studies
33. Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety.
34. Any contraindications against amivantamab (stages 1 and 2), carboplatin or pemetrexed (stage 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of one cycle of preoperative amivantamab therapy | 28 days pre-operative treatment
  The primary objective of this study is to determine the feasibility of four weeks of preoperative antibody therapy with amivantamab. Amivantamab will be administered as monotherapy (stage 1), and combined with carboplatin/pemetrexed chemotherapy (stage 2). Study treatment is followed by standard of care surgery, and (if clinically indicated) standard of care adjuvant therapy (chemotherapy, radiotherapy, EGFR tyrosine kinase inhibitor therapy) in patients with early stage or locally advanced non-small-cell lung cancer harboring oncogenic EGFR mutations who are eligible for curative resection.

SECONDARY OUTCOMES:
Characterization of residual tumor cells (if present) and immune cell infiltrate in resected tumors and lymph nodes | through study completion, an average of 1 year
  Secondary objectives are to characterize residual tumor cells (if present) and the immune cell infiltrate in resected tumors and lymph nodes following preoperative treatment with amivantamab (stage 1), and amivantamab plus carboplatin/pemetrexed (stage 2).

OTHER OUTCOMES:
ypTNM classification | immediately after the intervention/procedure/surgery
  Estimation of pathological tumor response rate per ypTNM classification and per IASLC recommendations (rate of complete pathological responses defined as absence of viable tumor cells on routine hematoxylin and eosin staining of resected tumors and lymph nodes; rate of major pathological responses defined as 10% or less viable tumor cells on routine hematoxylin and eosin staining of resected tumors)
R0 resection rate | immediately after the intervention/procedure/surgery
  Estimation of curative (R0) resection rate
RECIST assessment | immediately after the intervention/procedure/surgery and at12 months follow-up
  Assessment of radiologic response on preoperative computed tomography per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 Assessment of disease-free survival rate at 12 months per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Overall survival rate | through study completion, an average of 1 year
  Assessment of overall survival rate at 12 months; extended follow-up will be obtained within standard of care
Safety and tolerability of preoperative therapy with amivantamab | through study completion, an average of 1 year
  Assessment of safety and tolerability of preoperative therapy with amivantamab.
  Number (n) and percent (n/N) of AEs as assessed by CTCAE v5.0 Number of subjects (n) with at least one AE as assessed by CTCAE v5.0 Number (n) of SAEs as assessed by CTCAE v5.0 Number of subjects (n) with at least one SAE as assessed by CTCAE v5.0 Number of subjects (n) with AE related to Amivantamab treatment Number of subjects (n) with AE related to Chemotherapy treatment
  Events of special interests (ESIs):
  Number (n) of Infusion related reactions (IRRs) grade 3 or higher Number (n) of Interstitial Lung Disease/Pneumonitis Number (n) of Hepativ events (DILI or lab criteria (ALT/AST >= 5x ULN for 2 weeks or ALT/AST > 8x ULN, ALT/AST >=3x ULN if associated with the appearance or worsening of symptoms of liver injury, Persistens elevation or ALT/AST >=3x ULN for >=4 weeks)) Number (n) of subjects with at least one ESI
Estimation of morbidity and mortality within 90 days of surgery | Within 90 days after surgery
  Estimation of morbidity and mortality within 90 days of surgery
Exploratory translational parameters | through study completion, an average of 1 year
  Assessment of exploratory translational parameters in pretherapeutic samples and biopsies and resected tumor and lymph node samples, and blood cells, circulating nucleic acids, plasma, and serum withdrawn at several time points.
  Variant allele frequency of the dominant oncogenic EGFR mutation in percent [%] Quantitative analysis of CD68-positive macrophage in percent [%] Quantitative analysis of CD163-positive macrophages in percent [%] Quantitative analysis of CD56-positive natural killer cells in percent [%] Quantitative analysis of CD4-positive T lymphocytes in percent [%] Quantitative analysis of CD8-positive T lymphocytesin percent [%]
Exploratory translational parameters | through study completion, an average of 1 year
  Assessment of exploratory translational parameters in pretherapeutic samples and biopsies and resected tumor and lymph node samples, and blood cells, circulating nucleic acids, plasma, and serum withdrawn at several time points.

CONTACTS AND LOCATIONS:
Locations (4):
- Jessa Ziekenhuis, Department of Pneumology, Hasselt, Belgium
- Germany (2):
  - Thoraxklinik Heidelberg gGmbH, Studienzentrum Thoraxonkologie, Heidelberg, Baden-Wurttemberg
  - West German Cancer Center, Department of Medical Oncology, University Hospital Essen, Essen, Germany
- Erasmus Universitair Medisch Centrum Rotterdam Department of Pulmonary Medicine, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No